CLINICAL TRIAL: NCT04756310
Title: A Randomized, Multicenter Interventional Study of Nutritional Supplementation in Patients With Unilateral Wet AMD
Brief Title: Study of Nutritional Supplementation in Patients With Unilateral Wet AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Thea, Spain (Industry)
Collaborators: Alpha Bioresearch S.L. (Other); Investigación Estadística (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THEA_UNAV_1/14
Record Dates: First submitted 2015-12-04; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Wet Macular Degeneration
Keywords: AMD; Food Supplement; Antioxidant effect; Antiangiogenic effect; resveratrol
MeSH Terms: conditions — Wet Macular Degeneration | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Patients receiving Theavit food supplement considered as a placebo treatment for AMD condition.
  Two capsules/day before breakfast each day for 2 years
  Interventions: Dietary Supplement: Theavit
- Retilut (Experimental): Patients receiving Retilut food supplement. Two capsules/day before breakfast each day for 2 years
  Interventions: Dietary Supplement: Retilut

INTERVENTIONS:
Dietary Supplement: Retilut — antioxidants, antiangiogenic, antiinflammatory micronutrients
  Arms: Retilut
Dietary Supplement: Theavit — antioxidants micronutrients
  Other Names: food supplement
  Arms: Control

SUMMARY:
Retinal diseases are currently the leading cause of legal blindness in the developed world. Among these disorders, age-related macular degeneration (AMD) is one of the most prevalent conditions in individuals over 55 years of age. Late AMD, the most severe presentation of the disease, clinically manifests as either geographic atrophy (dry form) or choroidal neovascularization (CNV) (wet form). Although patients with wet AMD only represent 10% of the total cases, CNV is the main and most serious cause of central vision loss. At present, the treatment of wet AMD comprises intraocular injections of certain antiangiogenic agents which act by blocking VEGF (vascular endothelial growth factor). No effective treatment is yet available for dry AMD, though the AREDS (Age-Related Eye Disease Study) has shown that the administration of antioxidant supplements is able to slow progression of the disease. Such vitamin supplements are also indicated in patients who already have severe AMD (both exudative and atrophic) in one eye, since the risk of progression in these cases is high.

Recent studies involving new antioxidant and antiangiogenic molecules such as resveratrol, present in grapes and wine, have also revealed great efficacy in slowing the progression of advanced AMD. Hydroxytyrosol is another polyphenol with important antioxidant and antiinflammatory effects in the RPE.

Considering the above, the present randomized, multicenter interventional study involving Spanish and Portuguese patients with unilateral wet AMD was designed to compare the effects of two different nutritional supplements: one containing the antioxidants and minerals recommended by the AREDS at doses that can be used in the European Union (Theavit), and the other comprising these same substances plus omega-3 fatty acids (lipidic antioxidant), lutein (pigment protecting against light-induced damage) and resveratrol (antioxidant and antiangiogenic agent) (Retilut).

DETAILED DESCRIPTION:
Retinal diseases are currently the leading cause of legal blindness in the developed world. Among these disorders, age-related macular degeneration (AMD) is one of the most prevalent conditions in individuals over 55 years of age. In the United States, the prevalence of AMD varies from 0.5% at 55 years to 7% in people over 75 years. These data are clearly a cause for concern, in view of the aging of the population in developed countries. In Spain, a country with one of the greatest population aging problems, AMD affects 1.7% of all people over 50 years, and the incidence increases with age, reaching 18.5% among those over 85 years. AMD is characterized by progressive destruction of the central region of the retina (macula), resulting in central vision loss. While this does not lead to complete blindness, the associated impairment of autonomy has a very strong impact upon patient quality of life. AMD is a multifactorial disease - a fact that makes it difficult to establish the underlying etiology. In this sense, although only age is accepted as the principal factor associated to the development of AMD, other factors such as smoking, diet, oxidative stress, arterial hypertension or obesity have been extensively investigated in the context of the disease.

Late AMD, the most severe presentation of the disease, clinically manifests as either geographic atrophy (dry form) or choroidal neovascularization (CNV) (wet form). Although patients with wet AMD only represent 10% of the total cases, CNV is the main and most serious cause of central vision loss. At present, the treatment of wet AMD comprises intraocular injections of certain antiangiogenic agents such as ranibizumab, bevacizumab, aflibercept, etc., which act by blocking vascular endothelial growth factor (VEGF). No effective treatment is yet available for dry AMD, though the Age-Related Eye Disease Study (AREDS) has shown that the administration of antioxidant supplements is able to slow progression of the disease. Such vitamin supplements are also indicated in patients who already have severe AMD (both exudative and atrophic) in one eye, since the risk of progression in these cases is high.

The AREDS, sponsored by the National Eye Institute, was started in 1998 with the purpose of evaluating the effect of high-dose antioxidants (vitamins C and E, and beta-carotene) and minerals (zinc) upon the course of the disease. The results of the study showed that high levels of antioxidants and zinc significantly reduced the risk of progression towards advanced stages of AMD by 25%, and of vision loss by 19%. However, due to safety reasons, the doses used in the AREDS cannot be administered in the European Union, since they exceed the Recommended Daily Allowances (RDA). Therefore, the standard clinical practice is to use these substances in patients with high risk AMD as nutritional supplements at the usual RDAs. However, no interventional studies demonstrating the effects of these supplements have been carried out.

Following publication of the AREDS I, certain dietary intake studies suggested the importance of other molecules such as omega-3 fatty acids (DHA, EPA, DPA) and lutein / zeaxanthin. The AREDS work group therefore decided to conduct a new study including both nutrients in addition to those already evaluated (antioxidants and zinc). Lutein exerts an antioxidative effect, can act as a blue light filter, and moreover has antiinflammatory properties. This latter effect is especially important, considering that AMD is a disease secondary to a low-grade chronic inflammatory process of the retinal pigment epithelium (RPE). In addition to their antioxidant and antiinflammatory effects, the omega-3 fatty acids have important antiangiogenic properties, as evidenced both by in vitro and in vivo studies.

Recent studies involving new antioxidant and antiangiogenic molecules such as resveratrol, present in grapes and wine, have also revealed great efficacy in slowing the progression of advanced AMD. Hydroxytyrosol is another polyphenol with important antioxidant and antiinflammatory effects in the RPE.

Considering the above, the present randomized, multicenter interventional study involving Spanish and Portuguese patients with unilateral wet AMD was designed to compare the effects of two different nutritional supplements: one containing the antioxidants and minerals recommended by the AREDS at doses that can be used in the European Union (Theavit), and the other comprising these same substances plus omega-3 fatty acids (lipidic antioxidant), lutein (pigment protecting against light-induced damage) and resveratrol (antioxidant and antiangiogenic agent) (Retilut).

Study Design: A randomized, double-blind, multicenter interventional nutritional dose study was designed. The patient follow-up period will last 24 months. The estimated patient enrollment period will cover 9 months, and analysis of the results will be completed four months after the end of the follow-up period. The estimated total duration of the project will be between 52 months.

Study Subjects:

These patients from the different Spanish populations will be enrolled making use of the infrastructure afforded by the RETICS network, "Eye disease related to aging, vision quality and quality of life" (RD07/0062 subproject Retina). All patients will be 50 years old or more, and written informed consent will be obtained in all cases, together with authorization to enter their data in a database (data protection consent following the criteria of the Ethics Committees of each of the participating centers).

On the baseline visit, the patients will undergo a complete ophthalmological evaluation, and plasma will be collected for posterior analysis of several biochemical parameters.

Those patients who meet the inclusion criteria and none of the exclusion criteria will start nutritional supplementation for two years (2 daily capsule, nutritional dose) with one of the nutritional supplements. The study will be carried out on a simple-blind basis, even the patient knows the origin of the treatment, the ophthalmologist conducting follow-up will not know the composition of the provided supplement. Accordingly, the boxes and capsules will be adequately masked. The blisters with the nutritional supplements will be delivered to each patient at the inclusión visit (Day 0), and the empty blisters are to be returned as an initial measure of treatment compliance. Patient follow-up will take place every 6 months (Day 0, Month 6, Month 12, Month 18, Month 24), and will comprise a complete ophthalmological evaluation, with the registry of any ophthalmological adverse events. The appearance of such adverse events will be a secondary study endpoint, and is defined as the appearance of choroidal neovascularization in the fellow eye. First objective will be the measure of the change in the best corrected visual acuity (BCVA) in the study eye. Blood samples will be collected at Day 0, Month 12 and Month 24 for biochemical analysis (Luminex® markers, omega 3, lutein and zeaxanthin profile and plasma REDOX status) representing also a secondary study endpoints.

Ophthalmological examination:

* Visual acuity will be determined with the ETDRS system at a distance of four meters with the best optic correction.
* Anterior segment biomicroscopy study to discard opacification of the media. -Biomicroscopic funduscopy with +78/+90D lens.
* Digital retinography of the ocular fundus, red-free light photography of the fundus, and autofluorescence photography of the fundus under maximum pharmacologic mydriasis to ensure maximum image quality; a minimum of three examinations with photographs at 30/35° will be obtained.
* The follow-up of neovascularization will be carried out by fluorescein angiography and optical coherence tomography (OCT). The presence of subretinal and/or intraretinal fluid will be taken as a sign of wet AMD in OCT.

Biochemical analysis:

The plasma of the patients both on Day 0 and at the end of the study will be subjected to the following determinations:

* Analysis of the lipid profile (omega 3).
* Evaluation of the systemic oxidative condition based on total antioxidant capacity assay.
* Determination of lutein levels by HPLC.
* Detection of the main inflammatory and oxidative stress markers and/or vascular factors in plasma, based on Luminex® technology (affymetrix): VEGF-A, IL-1 beta, IL-6, IL-8, Eotaxin-2 (CCL24), HGF, PDGF, MCP-1, TNF-alpha and FGF.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥ 50 years.
2. Presence of unilateral choroidal neovascularisation or any of its clinical manifestations, such as disciform scars, subretinal hemorrhage, retinal pigment epithelium detachment associated to subretinal fluid and/or subretinal hemorrhage (stage V of the modified AREDS classification; AREDS, J.M. Seddon; IOVS 2009).
3. Patients who understand the conditions and particularities of the study and have given their written informed consent to participation in the trial.

Exclusion Criteria:

1. Patients with myopia > 6 dioptres.
2. Presence of posterior pole anomalies which can give rise to choroidal neovascularisation: nevi, angioid streaks, central serous choroidopathy, heredodegenerative retinal diseases, myopic choroidosis, diabetic retinopathy and choroiditis.
3. Media opacification precluding adequate assessment of the ocular fundus.
4. Patients who in the opinion of the investigator are very likely to not be able or not want to continue participating in the study.
5. Women of child-bearing potential who do not use a medically acceptable and highly effective contraceptive method (i.e., hormone implants, oral or parenteral contraceptives, together with condoms, certain intrauterine devices) from the inclusion visit and throughout the study treatment periods, up until two weeks after the study. Postmenopausal women (two years without menstruation) require no contraceptive method.
6. Patients having participated in any other treatment efficacy protocol in the previous three months.
7. Patients who will be participating in any other treatment efficacy protocol concomitant to the present study.
8. Patients using any type of nutritional supplement in the month before the screening visit.
9. Suspected or confirmed illegal drug abuse.
10. Incapacity of the patient and/or relatives to understand the study procedures, and thus inability to give informed consent.
11. Non-compliers, i.e., patients who fail to report to the follow-up visits or whose life style interferes with the protocol.
12. Patients under legal custody.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Best correct visual acuity (BCVA) | Comparison will be made of best visual acuity recorded in Month 12 versus that recorded on the baseline visit (Day 0).
  Variation in BCVA in the studied eye.
Best correct visual acuity (BCVA) | Comparison will be made of best visual acuity recorded in Month 24 versus that recorded on the baseline visit (Day 0).
  Variation in BCVA in the studied eye.

SECONDARY OUTCOMES:
Inflammatory markers | Determination will be made of the mean values obtained on visits Month 12 with respect to the recorded baseline values on visit Day 0
  VEGF-A, IL-1 beta, IL-6, IL-8, Eotaxin-2 (CCL24), HGF, PDGF, MCP-1, TNF-alfa and FGF.
Lipid blood profile | Determination will be made of the mean values obtained on visits Month 12 with respect to the recorded baseline values on visit Day 0
  Biochemical blood profile: Omega-3 lipid profile
Lipid blood profile | Determination will be made of the mean values obtained on visits Month 24 with respect to the recorded baseline values on visit Day 0
  Biochemical blood profile: Omega-3 lipid profile
Carotenoid profile | Determination will be made of the mean values obtained on visits Month 12 with respect to the recorded baseline values on visit Day 0
  Biochemical blood profile: lutein and zeaxantine values
Carotenoid profile | Determination will be made of the mean values obtained on visits Month 24 with respect to the recorded baseline values on visit Day 0
  Biochemical blood profile: lutein and zeaxantine values
Adverse Events | The percentage of these events will be the cumulative value on visits Month 6 in the study treatment group versus the control group.
  Determination and classification of simple and serious adverse events related or not to the study treatment and which appear in the contralateral eye.
Adverse Events | The percentage of these events will be the cumulative value on visits Month 12 in the study treatment group versus the control group.
  Determination and classification of simple and serious adverse events related or not to the study treatment and which appear in the contralateral eye.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo García-Layana, MD, Study Director — Clínica Universidad de Navarra; Roberto Gallego-Pinazo, MD, Principal Investigator — Hospital Universitario Politécnico La Fe; Emiliano Hernández-Galilea, MD, Principal Investigator — University of Salamanca; Miguel Ángel Zapata-Victori, MD, Principal Investigator — Hospital Universitario Vall d´Hebron; Maximino Abraldes, MD, PhD, Principal Investigator — Complexo Hospitalario Universitario de Santiago de Compostela; Rufino Silva, MD, PhD,FEBO, Study Director — Association for Innovation and Biomedical Research on Light and Image; Joao Nascimento, MD, Principal Investigator — Instituto de Retina e Diabetes Ocular de Lisboa; Jose J Escobar-Barranco, MD, Principal Investigator — Hospital Dos de Maig; Pilar Calvo, Md, PhD, Principal Investigator — Miguel Servet University Hospital, Zaragoza
Locations (9):
- Portugal (2):
  - AIBILI, Celas, Coimbra District
  - Instituto de Retina e Diabetes Ocular de Lisboa (IRL), Lisbon
- Spain (7):
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Miguel Servet University Hospital, Zaragoza, Aragon
  - Hospital Dos de Maig, Barcelona, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d´Hebrón, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Policlínico Universitario La Fe, Valencia